CLINICAL TRIAL: NCT03278522
Title: Comparison of Ramosetron Pre-treatment Time for Postoperative Nausea and Vomiting (PONV) and QTc Prolongation
Brief Title: Ramosetron Pre-treatment for PONV and QT Prolongation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Ka Young Rhee, Associate Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KUH1160112
Record Dates: First submitted 2017-09-06; First posted 2017-09-11 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: PONV; Prolonged QTc Interval
Keywords: ramosetron
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — ramosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ramosetron iv at induction (I) (Active Comparator): 0.6mg of ramosetron is given to the patients intravenously at anesthesia induction
  Interventions: Drug: Ramosetron
- ramosetron iv at recovery (R) (Active Comparator): 0.6mg of ramosetron is given to the patients intravenously at end of surgery
  Interventions: Drug: Ramosetron

INTERVENTIONS:
Drug: Ramosetron — Intravenous ramosetron 0.6mg is given to the patients at the induction of anesthesia, or at the end of surgery
  Other Names: ramosetron pre-treatment

SUMMARY:
Ramosetron is commonly used to prevent postoperative nausea and vomiting (PONV) in the Eastern Asia. The prolongation of QTc interval is a main side effect. In this study, the pre-treatment time of ramosetron to decrease PONV, and QTc prolongation is compared.

DETAILED DESCRIPTION:
This prospective study evaluate 42 female patients who underwent laparoscopic gynecologic surgery under general anesthesia. Group I (n=21) receive 0.6mg of ramosetron at anesthesia induction. Group R (n=21) received the same at the end of surgery. PONV is evaluated at arrival to post-anesthetic care unit (PACU), before induction, discharge from PACU, 24-, 48-, and 72- after discharge from PACU. The QTc interval is checked before anesthesia, at arrival to PACU, and 24-h after discharge from PACU.

Forty two subjects are needed with an α value of 0.05, a power of 0.8, and effect size difference of 0.9.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent laparoscopic gynecologic surgery

Exclusion Criteria:

* preoperative bradyarrhythmia in ECG

Ages: 19 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
QTc interval change | within 10 min after arrival at PACU, and 24 hour after discharge from PACU
  Difference of QTc interval from preoperative value

CONTACTS AND LOCATIONS:
Overall Officials: Ka Young Rhee, MD,PhD, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Lee Sung Ho, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided